CLINICAL TRIAL: NCT04101058
Title: Treatment Response Among Chinese Patients With Acute Attack of Neuromyelitis Optica Spectrum Disorders: A Prospective, Multicenter Real-world Study
Brief Title: Treatment Response Among Chinese Neuromyelitis Optica Spectrum Disorders
Acronym: Momentum
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guangdong 999 Brain Hospital (Other)
Responsible Party: Principal Investigator, Wei Qiu, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 201809
Record Dates: First submitted 2018-12-14; First posted 2019-09-24 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuromyelitis Optica (NMO)/ Neuromyelitis Optica Spectrum Disorders (NMOSD) is an immune-mediated inflammatory demyelinating disease of the central nervous system mainly involving optic nerve and spinal cord. It is clinically characterized by simultaneous or sequential involvement of the optic nerve and spinal cord, presenting a progressive or remission and relapse course, which can lead to paralysis and blindness.

The objective of this study is to provide evidence regarding treat effects and factors related to prognosis which will help physicians better evaluable risk-benefit in NMOSD management and improve patients' outcome.

DETAILED DESCRIPTION:
Neuromyelitis Optica (NMO)/ Neuromyelitis Optica Spectrum Disorders (NMOSD) is an immune-mediated inflammatory demyelinating disease of the central nervous system mainly involving optic nerve and spinal cord. It is clinically characterized by simultaneous or sequential involvement of the optic nerve and spinal cord, presenting a progressive or remission and relapse course, which can lead to paralysis and blindness.

Globally, there is no solid data available for the diagnosis, treatment and prognosis of patients with acute Neuromyelitis Optica Spectrum Disorders (NMOSD) attack, particularly very rare data from prospective studies. This is a multicenter, prospective, real-world cohort study in patients with acute NMOSD attack in China.

Baseline data for approximately 200 patients with acute NMOSD attack from approximately 4 centers will be collected. Patients with acute NMOSD attack (including first episodes and relapses) whose expansile disability status score (EDSS ) ≥ 2 points at baseline will be eligible to be further included in prospective study cohort for analysis of treatment effects and prognosis.

The objective of this study is to provide evidence regarding treat effects and factors related to prognosis which will help physicians better evaluable risk-benefit in NMOSD management and improve patients' outcome.

ELIGIBILITY:
1. Inclusion criteria for patients with baseline data collection:

1. The subject can fully understand the content of the study and voluntarily sign the informed consent form;
2. Male or female ≥18 years old;
3. Diagnosed as NMOSD based on 2015 NMOSD diagnostic criteria of International NMO Diagnostic Team (IPND) and currently under acute attack.

2. Inclusion criteria for subjects enrolled in a prospective study cohort should further meet:

1. The subject can fully understand the content of the study and voluntarily sign the informed consent form;
2. Male or female,≥18 years old;
3. Diagnosed as NMOSD based on 2015 NMOSD diagnostic criteria of International NMO Diagnostic Team (IPND) and currently under acute attack.
4. Subjects with acute attack (including first episodes and relapse) should have an EDSS of ≥ 2 at baseline; and for patients with acute relapse, new symptoms or the primary symptoms, being judged by investigator, should have been aggravated for 24 hours or more [11-13];
5. The subject should have typical symptoms of movement, sensation, vision, defecation/urination or nausea/vomiting at attack;
6. Subjects should agree to participate in the study, and to receive AQP4-IgG examination before and after treatment;
7. Subjects should agree to undergo an ophthalmologic examination before and after treatment;
8. Subjects should agree to participate the study and agree to have the collected data analyzed by this study.

3. Exclusion criteria:

1. Subjects treated with study medication in another clinical trial during the last 30 days or 5 half-life periods prior to screening or during the effect period of the drug, whichever is the longest; Note: Subjects who participated in an observational study (ie, the study did not require changes to medication or other interventions) were not excluded.
2. Immediate relatives of the researcher/research center staff directly related to the study, or the researcher/research center staff directly related to the study ("immediate relatives" refer to spouses, parents, children or siblings (Whether it's biological or legal adoption).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute episode of Neuromyelitis Optica Spectrum Disorders (NMOSD)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Expansile Disability Status Score | at the end of the first high-dose intravenous Methylprednisone (IVMP) therapy (up to 3 weeks )among subjects who received high-dose IVMP
  Compared with baseline, changes in EDSS（Expansile Disability Status Score ）at the end of the first high-dose intravenous Methylprednisone (IVMP) therapy among subjects who received high-dose IVMP.
  EDSS score is based on the evaluation of eight functional systems of the central nervous system.The total score of the assessment is between 0 and 10 points, and each 0.5 is divided into one grade, which is divided into 20 grades.

SECONDARY OUTCOMES:
Expansile Disability Status Score | at discharge (7 days after last treatment)
  Compared with baseline, proportion of subjects with EDSS improved ≥1 point at discharge (7 days after last treatment)
Changes In AQP4-IgG | at the end of the first IVMP therapy（up to 3 weeks) among subjects who received high-dose IVMP
  Compared with baseline , changes in AQP4-IgG at the end of the first IVMP therapy among subjects who received high-dose IVMP
As Assessed By Snellen Chart | at the end of the first high-dose IVMP theraty (up to 3 weeks) among subjects who received high-dose IVMP
  Compared with baseline , changes in visual acuity (as assessed by Snellen chart) at the end of the first high-dose IVMP therapy among subjects who received high-dose IVMP
PGI-I Score | at the end of the first high-dose IVMP therapy(up to 3 weeks) among subjects who received high-dose IVMP
  Score of Patient Global Improvement-Impression (PGI-I) at the end of the first high-dose IVMP therapy among subjects who received high-dose IVMP Patient Global Impressions (PGI)-Improvement Mark the box that best describes how you (the patient) have felt in general since you started taking this medicine. (Choose one)
  1 = Very assessed, 2 = Much better, 3 = A little better, 4 = The same, 5 = A little worse, 6 = Much worse, 7 = Very much worse
Changes In AQP4-IgG | at discharge (7 days after the last treatment)
  Compared with baseline , changes in AQP4-IgG at discharge (7 days after the last treatment) * among subjects who received high-dose IVMP
As Assessed By Snellen Chart | at discharge (7 days after the last treatment)
  Compared with baseline, changes in visual acuity (as assessed by Snellen chart) at discharge (7 days after the last treatment)* among subjects who received high-dose IVMP
PGI-I Score | at discharge (7 days after the last treatment)
  Score of Patient Global Improvement-Impression (PGI-I) at discharge (7 days after the last treatment)* among subjects who received high-dose IVMP
Expansile Disability Status Score | at discharge (7 days after the last treatment)
  Compared with baseline, changes in EDSS at discharge (7 days after the last treatment) * among subjects who received high-dose IVMP
The proportion of patients who did not respond to the first high-dose IVMP therapy(up to 3 weeks) | at discharge (7 days after the last treatment)
  The proportion of patients who did not respond to the first high-dose IVMP therapy(up to 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Qiu, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Wei Qiu, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papadopoulos MC, Bennett JL, Verkman AS. Treatment of neuromyelitis optica: state-of-the-art and emerging therapies. Nat Rev Neurol. 2014 Sep;10(9):493-506. doi: 10.1038/nrneurol.2014.141. Epub 2014 Aug 12. PMID 25112508
- [Background] Lennon VA, Kryzer TJ, Pittock SJ, Verkman AS, Hinson SR. IgG marker of optic-spinal multiple sclerosis binds to the aquaporin-4 water channel. J Exp Med. 2005 Aug 15;202(4):473-7. doi: 10.1084/jem.20050304. Epub 2005 Aug 8. PMID 16087714
- [Background] Kim SH, Kim W, Li XF, Jung IJ, Kim HJ. Repeated treatment with rituximab based on the assessment of peripheral circulating memory B cells in patients with relapsing neuromyelitis optica over 2 years. Arch Neurol. 2011 Nov;68(11):1412-20. doi: 10.1001/archneurol.2011.154. Epub 2011 Jul 11. PMID 21747007
- [Background] Bizzoco E, Lolli F, Repice AM, Hakiki B, Falcini M, Barilaro A, Taiuti R, Siracusa G, Amato MP, Biagioli T, Lori S, Moretti M, Vinattieri A, Nencini P, Massacesi L, Mata S. Prevalence of neuromyelitis optica spectrum disorder and phenotype distribution. J Neurol. 2009 Nov;256(11):1891-8. doi: 10.1007/s00415-009-5171-x. Epub 2009 May 28. PMID 19479168
- [Background] Kawachi I, Lassmann H. Neurodegeneration in multiple sclerosis and neuromyelitis optica. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):137-145. doi: 10.1136/jnnp-2016-313300. Epub 2016 Sep 26. PMID 27671902
- [Background] Pandit L, Asgari N, Apiwattanakul M, Palace J, Paul F, Leite MI, Kleiter I, Chitnis T; GJCF International Clinical Consortium & Biorepository for Neuromyelitis Optica. Demographic and clinical features of neuromyelitis optica: A review. Mult Scler. 2015 Jun;21(7):845-53. doi: 10.1177/1352458515572406. Epub 2015 Apr 28. PMID 25921037
- [Background] Optic Neuritis Study Group. Multiple sclerosis risk after optic neuritis: final optic neuritis treatment trial follow-up. Arch Neurol. 2008 Jun;65(6):727-32. doi: 10.1001/archneur.65.6.727. PMID 18541792
- [Background] Weinshenker BG, O'Brien PC, Petterson TM, Noseworthy JH, Lucchinetti CF, Dodick DW, Pineda AA, Stevens LN, Rodriguez M. A randomized trial of plasma exchange in acute central nervous system inflammatory demyelinating disease. Ann Neurol. 1999 Dec;46(6):878-86. doi: 10.1002/1531-8249(199912)46:63.0.co;2-q. PMID 10589540
- [Background] Kim SH, Kim W, Huh SY, Lee KY, Jung IJ, Kim HJ. Clinical efficacy of plasmapheresis in patients with neuromyelitis optica spectrum disorder and effects on circulating anti-aquaporin-4 antibody levels. J Clin Neurol. 2013 Jan;9(1):36-42. doi: 10.3988/jcn.2013.9.1.36. Epub 2013 Jan 3. PMID 23346159
- [Background] Wingerchuk DM, Banwell B, Bennett JL, Cabre P, Carroll W, Chitnis T, de Seze J, Fujihara K, Greenberg B, Jacob A, Jarius S, Lana-Peixoto M, Levy M, Simon JH, Tenembaum S, Traboulsee AL, Waters P, Wellik KE, Weinshenker BG; International Panel for NMO Diagnosis. International consensus diagnostic criteria for neuromyelitis optica spectrum disorders. Neurology. 2015 Jul 14;85(2):177-89. doi: 10.1212/WNL.0000000000001729. Epub 2015 Jun 19. PMID 26092914
- [Background] Araki M, Matsuoka T, Miyamoto K, Kusunoki S, Okamoto T, Murata M, Miyake S, Aranami T, Yamamura T. Efficacy of the anti-IL-6 receptor antibody tocilizumab in neuromyelitis optica: a pilot study. Neurology. 2014 Apr 15;82(15):1302-6. doi: 10.1212/WNL.0000000000000317. Epub 2014 Mar 14. PMID 24634453
- [Background] Yamasaki R, Matsushita T, Fukazawa T, Yokoyama K, Fujihara K, Ogino M, Yokota T, Miyamoto K, Niino M, Nomura K, Tomioka R, Tanaka M, Kawachi I, Ohashi T, Kaida K, Matsui M, Nakatsuji Y, Ochi H, Fukaura H, Kanda T, Nagaishi A, Togo K, Mizusawa H, Murai H, Kira J. Efficacy of intravenous methylprednisolone pulse therapy in patients with multiple sclerosis and neuromyelitis optica. Mult Scler. 2016 Sep;22(10):1337-48. doi: 10.1177/1352458515617248. Epub 2015 Nov 12. PMID 26564994
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] van Winsen LM, Polman CH, Dijkstra CD, Tilders FJ, Uitdehaag BM. Suppressive effect of glucocorticoids on TNF-alpha production is associated with their clinical effect in multiple sclerosis. Mult Scler. 2010 Apr;16(4):500-2. doi: 10.1177/1352458509359721. Epub 2010 Jan 19. PMID 20086025
- [Background] Abboud H, Petrak A, Mealy M, Sasidharan S, Siddique L, Levy M. Treatment of acute relapses in neuromyelitis optica: Steroids alone versus steroids plus plasma exchange. Mult Scler. 2016 Feb;22(2):185-92. doi: 10.1177/1352458515581438. Epub 2015 Apr 28. PMID 25921047
- [Background] Holladay JT. Visual acuity measurements. J Cataract Refract Surg. 2004 Feb;30(2):287-90. doi: 10.1016/j.jcrs.2004.01.014. No abstract available. PMID 15030802
- [Derived] Wang J, Cui C, Lu Y, Chang Y, Wang Y, Li R, Shan Y, Sun X, Long Y, Wang H, Wang Z, Lee M, He S, Lu Z, Qiu W, Tan S. Therapeutic Response and Possible Biomarkers in Acute Attacks of Neuromyelitis Optica Spectrum Disorders: A Prospective Observational Study. Front Immunol. 2021 Aug 4;12:720907. doi: 10.3389/fimmu.2021.720907. eCollection 2021. PMID 34421925